CLINICAL TRIAL: NCT03517722
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study of Ustekinumab in Subjects With Active Systemic Lupus Erythematosus
Brief Title: A Study of Ustekinumab in Participants With Active Systemic Lupus Erythematosus
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated early as a result of the outcome of the pre-planned Interim Analysis
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108440; 2017-001489-53 (EudraCT Number); CNTO1275SLE3001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2018-04-13; First posted 2018-05-07 (Actual); Results first posted 2022-03-09 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Lupus Erythematosus, Systemic
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ustekinumab (Experimental): Participants will receive ustekinumab approximately 6 milligram per kilogram (mg/kg) intravenously (IV) based on body weight-range at Week 0 followed by 90 mg ustekinumab subcutaneously (SC) at Week 8 and every 8 weeks (q8w) thereafter through Week 48 during double-blind period. Eligible participants who will enter the extension period will continue to receive 90 mg ustekinumab SC q8w through Week 160.
  Interventions: Drug: Ustekinumab (approximately 6 mg/kg); Drug: Ustekinumab 90 mg
- Placebo (Experimental): Participants will receive matching placebo to ustekinumab IV at Week 0, followed by matching placebo to ustekinumab SC at Week 8 and q8w thereafter through Week 48 during double-blind period. Eligible participants who will enter the extension period will cross-over to receive 90 mg ustekinumab SC q8w through Week 160.
  Interventions: Drug: Placebo; Drug: Ustekinumab 90 mg

INTERVENTIONS:
Drug: Placebo — Participants will receive placebo matching to ustekinumab IV or SC.
  Arms: Placebo
Drug: Ustekinumab (approximately 6 mg/kg) — Participants will receive ustekinumab approximately 6 mg/kg via IV route based on body weight-range.
  Other Names: Stelara
  Arms: Ustekinumab
Drug: Ustekinumab 90 mg — Participants will receive 90 mg ustekinumab via SC route.
  Other Names: Stelara

SUMMARY:
The purpose of this study is to evaluate the efficacy of ustekinumab in participants with active systemic lupus erythematosus (SLE) who have not adequately responded to one or more standard of care treatments.

DETAILED DESCRIPTION:
This study evaluates the efficacy, safety, and tolerability of ustekinumab in participants with active SLE according to Systemic Lupus International Collaborating Clinics (SLICC) criteria Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score greater than (>=) 6, despite receiving one or more standard-of-care treatments (example, immunomodulators, antimalarial drugs, and/or glucocorticoids). The total duration of the study is up to 182 weeks, consisting of 3 study periods: a screening period (approximately 6 weeks), a double blind period (52 weeks), and an extension period (124 weeks). Other study evaluations will include pharmacokinetics, immunogenicity, biomarkers and pharmacogenomic evaluations. The safety of the participants enrolled in the study will be monitored on an ongoing basis throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female
* Has a documented medical history (that is, met at least 1 of the two criteria below) that participant met the Systemic Lupus International Collaborating Clinics (SLICC) classification criteria for systemic lupus erythematosus (SLE) at least 3 months prior to first dose of study agent:

  1. Met a total of at least 4 SLICC criteria, including at least 1 clinical and at least 1 immunologic;
  2. Has a diagnosis of lupus nephritis, confirmed by renal biopsy and at least 1 of the following autoantibodies: antinuclear antibodies (ANA) or anti-double-stranded deoxyribonucleic acid (anti-dsDNA)
* Has a positive test in the medical history and confirmed at screening for at least 1 of the following autoantibodies: antinuclear antibodies, anti-double-stranded deoxyribonucleic acid, and/or anti-Smith
* Has greater than or equal to (>=) 1 British Isles Lupus Assessment Group (BILAG) A and/or >= 2 BILAG B scores observed during screening
* Has a Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) activity score >=4 (excluding diffuse non-inflammatory alopecia) or >= 4 joints with pain and signs of inflammation at screening, Week 0, or both
* Has a Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score >=6 at screening. Must also have SLEDAI-2K >= 4 for clinical features (excluding headache and laboratory abnormalities) at Week 0
* Cannot be pregnant, nursing, intending to become pregnant, or unwilling to follow contraception or egg/sperm donation guidelines
* Must be receiving stable doses of >=1 protocol-permitted standard of care SLE treatment: oral glucocorticoids, anti-malarials, immunomodulators (methotrexate, azathioprine, 6-mercaptopurine, mycophenolate mofetil, mycophenolic acid)

Exclusion Criteria:

* Has any unstable or progressive SLE manifestation (example: central nervous system lupus, systemic vasculitis, end-stage renal disease, severe or rapidly progressive glomerulonephritis, pulmonary hemorrhage, myocarditis) that may warrant escalation in therapy beyond permitted background medications. Participants requiring renal hemodialysis or peritoneal dialysis are also excluded
* Has other co-existent inflammatory diseases (example: rheumatoid arthritis, psoriasis, psoriatic arthritis, Crohn's disease)
* Has a urinary protein to creatinine ratio of greater than (>)4 gram per gram (g/g) per day
* Has an acute or chronic infectious illness (example: human immunodeficiency virus, hepatitis B or C virus, tuberculosis, opportunistic infections)
* Has a history of cancer or lymphoproliferative disease within the last 5 years except for treated and non-recurrent cutaneous basal cell carcinoma, squamous cell carcinoma, or cervical carcinoma
* Has any condition requiring multiple courses of systemic glucocorticoids (example: uncontrolled asthma, chronic obstructive pulmonary disease)
* Has a history of major surgery within the last month
* Has received live virus or bacterial vaccines within 16 weeks prior to first dose of study agent or Bacille Calmette-Guerin (BCG) vaccination within 12 months of screening
* Has previously received ustekinumab
* Has received cyclophosphamide orally within 90 days or intravenously within 180 days of screening
* Has received a single B-cell targeted therapy (e.g. belimumab) within 3 months, >1 previous B-cell targeted therapy within 6 months, or B-cell depleting therapy (example: rituximab) within 12 months of first dose of study agent
* Has received protocol-prohibited oral or biologic immunomodulatory therapy in the last 3 months or less than (<)5 half-lives (whichever is longer) prior to first dose of study agent
* Has received adrenocorticotropic hormone (ACTH) within 1 month prior to first dose of study agent
* Has received epidural, intravenous, intramuscular, intraarticular, intrabursal, intralesional glucocorticoids within 6 weeks of first dose of study agent
* Locally-delivered therapies except for ophthalmic use of cyclosporine A or topical use of nonsteroidal anti inflammatory drugs (NSAIDs), analgesics, or high-potency glucocorticoids (World Health Organization criteria) are prohibited

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 516 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2020-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (204):
- United States (69):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Achieve Clinical Research, LLC, Vestavia Hills, Alabama
  - Medvin Clinical Research, Covina, California
  - Lugene Eye Institute, Glendale, California
  - C.V. Mehta, MD Medical Corp., Hemet, California
  - University of California at San Diego, La Jolla, California
  - Advanced Medical Research - Lakewood, Lakewood, California
  - Loma Linda University, Loma Linda, California
  - Loma Linda University Health Care, Loma Linda, California
  - Valerius Medical Group & Research Center, Los Alamitos, California
  - Keck School of Medicine of USC, Los Angeles, California
  - Wallace Rheumatic Study Center, Los Angeles, California
  - East Bay Rheumatology Medical Group, San Leandro, California
  - Westlake Medical Research Clinical Trials, Thousand Oaks, California
  - University Clinical Investigators, Inc, Tustin, California
  - Inland Rheumatology Clinical Trials Inc., Upland, California
  - University of Colorado, Aurora, Colorado
  - Denver Arthritis Clinic, Denver, Colorado
  - UPMC Lupus Center of Excellence, New Haven, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Arthritis and Rheumatic Disease Specialties, Aventura, Florida
  - Bay Area Arthritis and Osteoporosis, Brandon, Florida
  - Centre for Rheumatology, Immunology and Arthritis, Fort Lauderdale, Florida
  - University of Florida Health Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Rheumatology Associates of Central Florida, PA, Orlando, Florida
  - Omega Research Consultants, Orlando, Florida
  - Millennium Research, Ormond Beach, Florida
  - Integral Rheumatology And Immunology Specialists, Plantation, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Piedmont Healthcare - Piedmont Hospital, Atlanta, Georgia
  - DeKalb Medical Specialty Center, Decatur, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Graves-Gilbert Clinic - Bowling Green, Bowling Green, Kentucky
  - Arthritis and Diabetes Clinic, Monroe, Louisiana
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - June DO, PC., Lansing, Michigan
  - St Paul Rheumatology PA, Eagan, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Oklahoma Medical Research Foundation, Las Vegas, Nevada
  - Innovative Health Research, Las Vegas, Nevada
  - Albuquerque Center for Rheumatology, Albuquerque, New Mexico
  - Biomedical Research Alliance Of New York, Lake Success, New York
  - The Feinstein Institute for Medical Research, Manhasset, New York
  - NYU Center for Musculoskeletal Care, New York, New York
  - Hospital for Special Surgery, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Joint and Muscle Research Institute, Charlotte, North Carolina
  - DJL Clinical Research, PLLC, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - OK Center for Arthritis Therapy & Research, Inc., Tulsa, Oklahoma
  - Lewis Katz School of Medicine, Temple University, Philadelphia, Pennsylvania
  - Allegheny Rheumatology/Allegheny Singer Research Institute, Wexford, Pennsylvania
  - Columbia Arthritis Center, Columbia, South Carolina
  - West Tennessee Research Institute, Jackson, Tennessee
  - Dr. Ramesh Gupta, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Amarillo Center for Clinical Research, Amarillo, Texas
  - Austin Regional Clinic, Austin, Texas
  - Arthritis Centers of Texas, Dallas, Texas
  - Sun Research Institute, San Antonio, Texas
  - UT Health Science Center at San Antonio, San Antonio, Texas
  - University of Washington, Seattle, Washington
  - Rheumatology and Pulmonary Clinic, Beckley, West Virginia
- Argentina (8):
  - Fundacion CENIT para la Investigacion en Neurociencias, Buenos Aires
  - Instituto Centenario, Buenos Aires
  - Centro Privado de Medicina Familiar, Buenos Aires
  - Framingham Centro Medico, Ciudad de La Plata
  - Hospital Escuela 'Gral. Jose F. de San Martin', Corrientes
  - Hospital Italiano de Cordoba, Córdoba
  - CER San Juan Centro Polivalente de Asistencia e Investigacion Clinica, San Juan
  - Centro Medico Privado de Reumatologia, San Miguel de Tucumán
- Bulgaria (4):
  - MHAT Trimantium, Plovdiv
  - Diagnostic-Consultative Center (DCC) Aleksandrovska, Sofia
  - UMHAT St. Ivan Rilski, Sofia
  - Medical Centre Synexus, Sofia
- Canada (5):
  - University of Calgary, Calgary, Alberta
  - University of Manitoba, Winnipeg, Manitoba
  - McMaster University, Hamilton, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - CHU de Québec, Québec, Quebec
- China (9):
  - The First Affiliated Hospital of Baotou Medical University, Baotou
  - Peking Union Medical College Hospital, Beijing
  - West China Hospital Sichuan University, Chengdu
  - Guangdong Provincial People's Hospital, Guangzhou
  - Affiliated Hospital of Inner Mongolia Med U, Hohhot
  - Shanghai Ruijin Hospital, Shanghai
  - Tianjin Medical University General Hospital, Tianjin
  - Tongji Hospital of Tongji Medical College of Huangzhong Univ, Wuhan
  - The 1st affiliated Hospital of Xi'an Traffic University, Xi'an
- Colombia (6):
  - Centro de Investigación en Reumatología y especialidades médicas S.A.S. - CIREEM S.A.S., Bogotá
  - IPS Medicity SAS, Bucaramanga
  - Servimed S A S, Bucaramanga
  - Preventive Care Ltda, Chía
  - Clinica Universitaria Bolivariana, Medellín
  - Funcentra, Montería
- Germany (5):
  - Charite - Universitaetsmedizin Berlin (CCM), Berlin
  - Medizinische Hochschule Hannover, Hanover
  - Rheumazentrum Ruhrgebiet, Herne
  - Rheumatology Unit, Leipzig
  - Universitaetsmedizin Mainz, Mainz
- Hungary (3):
  - Szt, Istvan and Szt. Laszlo, Budapest
  - Bekes Megyei Pandy Kalman Korhaz, Gyula
  - Belvarosi Egeszseghaz Kft. (Leda-Platan Maganklinika es Sebeszeti Kozpont), Zalaegerszeg
- Japan (22):
  - Chiba University Hospital, Chiba
  - National Hospital Organization Chiba East Hospital, Chiba
  - Hospital of the University of Occupational and Enviromental Health, Fukuoka
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Hiroshima Red Cross Hospital & Atomic-bomb Survivors Hospital, Hiroshima
  - National Hospital Organization Osaka Minami Medical Center, Kawachi-Nagano
  - Kawasaki Rheumatism and Internal Medicine Clinic, Kitakyushu
  - Toho University Medical Center, Ohashi Hospital, Meguro-ku
  - Nagasaki University Hospital, Nagasaki
  - National Hospital Organization Nagoya Medical Center, Nagoya
  - Kitasato University Hospital, Sagamihara
  - Sapporo City General Hospital, Sapporo
  - Hokkaido University Hospital, Sapporo
  - Sasebo Chuo Hospital, Sasebo
  - Tohoku University Hospital, Sendai
  - Keio University Hospital, Shinjuku-ku
  - Center Hospital of the National Center for Global Health and Medicine, Shinjuku-ku
  - St. Luke's International Hospital, Tokyo
  - Juntendo University Hospital, Tokyo
  - Fujita Health University Hospital, Toyoake
  - National Hospital Organization Yokohama Medical Center, Yokohama
- Lithuania (4):
  - Lietuvos sveikatos mokslų universiteto ligoninė Kauno klinik, Kaunas
  - Klaipeda University Hospital, Klaipėda
  - Vaiku ligonine Vilniaus Universiteto ligon. Santariskiu fil, Vilnius
  - Vilnius University Hospital Santariskiu Clinics, Vilnius
- Poland (10):
  - Szpital Uniwersytecki nr 2 im dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - Nzoz Bif Med, Bytom
  - Centrum Medyczne AMED oddzial w Lodzi, Lodz
  - Samodzielny Publiczny Szpital Kliniczny Nr 4 w Lublinie, Lublin
  - Twoja Przychodnia - Centrum Medyczne Nowa Sol, Nowa Sól
  - Centrum Medyczne Medens S.C. Grupowa Praktyka Lekarska, Sonoswiec
  - Centrum Medyczne Pratia Tychy, Tychy
  - Centrum Medyczne Pratia Warszawa, Warsaw
  - Reumatika-Centrum Reumatologii, NZOZ, Warsaw
  - Uniwersytecki Szpital Kliniczny im. J. Mikulicza-Radeckiego, Wroclaw
- Portugal (5):
  - Instituto Portugues de Reumatologia, Lisbon
  - Uls Sao Jose - Hosp. Curry Cabral, Lisbon
  - Hosp. Da Luz Lisboa, Lisbon
  - ULSAM, EPE - Hospital Conde de Bertiandos, Ponte de Lima
  - C.H. de Vila Nova de Gaia/Espinho, Vila Nova de Gaia
- Russia (8):
  - Regional Clinical Hospital for War Veterans, Kemerovo
  - LLL Medical Center Revma-Med, Kemerovo
  - Clinical Diagnostic Center 'Ultramed', Omsk
  - Northen-Western State Medical University n.a. I.I. Mechnikov, Saint Petersburg
  - Leningrad region clinical hospital, Saint Petersburg
  - City Clinical Hospital #31, Saint Petersburg
  - Ulyanovsk Regional Clinical Hospital, Ulyanovsk
  - Clinical Emergency Hospital n.a. N.V. Solovyev, Yaroslavl
- Serbia (7):
  - Institute of Rheumatology Belgrade, Belgrade
  - Institute of Rheumatology, Belgrade
  - Military Medical Academy, Belgrade
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - University Clinical Center Kragujevac, Kragujevac
  - Institute for Treatment and Rehabilitation Niska Banja, Niška Banja
  - Clinical Center of Vojvodina, Vojvodina
- South Africa (4):
  - Panorama Medical Centre, Cape Town
  - Excellentis Clinical trial Consultants, George
  - Clinical Research Unit, University of Pretoria, Pretoria
  - Winelands Medical Research Centre, Stellenbosch
- South Korea (5):
  - Daegu Catholic University Medical Center, Daegu
  - Chonbuk National Univ Hospital, Jeonju
  - Seoul National University Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Ajou University Hospital, Suwon
- Spain (9):
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Univ. de Basurto, Bilbao
  - Hosp Reina Sofia, Córdoba
  - Hosp. Clinico San Carlos, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp Regional Univ de Malaga, Málaga
  - Hosp. Univ. Infanta Sofia, San Sebastián de los Reyes
  - Hosp. Infanta Luisa, Seville
  - Hosp. Do Meixoeiro, Vigo -Pontevedra
- Taiwan (8):
  - Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital, Kwei-san Hsiang
  - Chung Shan Medical University Hospital, Taichung
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Cathay General Hospital, Taipei
  - Taipei Medical University, Taipei
  - Taipei Veterans General Hospital, Taipei
- Thailand (6):
  - Phramongkutklao Hospital and Medical College, Bangkok
  - Rajavhiti Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Songklanagarind hospital, Hat Yai
  - Chiang Mai University, Muang
- Ukraine (7):
  - Mechnikov Inst, Miska bagatoprofilna likarnia #18, Kharkiv
  - Kyiv City Clinical Hospital #3, Kyiv
  - Kyivska oblasna klinichna likarnia, Kyiv
  - Odeska oblasna klinichna likarnia, Odesa
  - Multidisciplinary Medical Center of Odessa National Medical University, Odesa
  - MNPE 'Vinnytsia Regional Clinical Hospital named after M.I. Pyrogov of Vinnytsia Regional Council', Vinnytsia
  - Naukovo-doslidnyi inst. Reabilit. Pyrogova [Revmatologichne], Vinnytsia

REFERENCES:
- [Derived] van Vollenhoven RF, Kalunian KC, Dorner T, Hahn BH, Tanaka Y, Gordon RM, Shu C, Fei K, Gao S, Seridi L, Gallagher P, Lo KH, Berry P, Zuraw QC. Phase 3, multicentre, randomised, placebo-controlled study evaluating the efficacy and safety of ustekinumab in patients with systemic lupus erythematosus. Ann Rheum Dis. 2022 Oct 12;81(11):1556-1563. doi: 10.1136/ard-2022-222858. PMID 35798534
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR108440&attachmentIdentifier=e67c0fcb-bac3-4351-a715-45375e8b9704&fileName=2017-001489-53___Receipt.png&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants received study drug up to Week 113, but were assessed for safety up to Week 130 (that is, after study termination).
Groups:
- Placebo to Ustekinumab: Participants received matching placebo to ustekinumab intravenously (IV) 6 milligrams per kilogram (mg/kg) based on body weight at Week 0 followed by matching placebo to ustekinumab subcutaneously (SC) 90 mg at Week 8 and every 8 weeks (q8w) thereafter through Week 48 during double-blind period. At Week 52, participants who entered the open-label extension period crossed over to receive ustekinumab 90 mg SC q8w through Week 113.
- Ustekinumab: Participants received ustekinumab 6 mg/kg IV based on body weight (ustekinumab 260 mg [weight less than or equal to {<=} 55 kg]; ustekinumab 390 mg [weight greater than {>} 55 kg and <= 85 kg] at Week 0 followed by ustekinumab 90 mg SC at Week 8 and q8w thereafter through Week 48 during double-blind period. At Week 52, participants who entered the open-label extension period continued to receive ustekinumab 90 mg SC q8w through Week 113.
Period: Double Blind Period: Week 0-52
Arm/Group | Placebo to Ustekinumab | Ustekinumab
Started | 208 | 308
Treated | 208 | 307
Completed | 105 | 153
Not Completed | 103 | 155
Not completed — Adverse Event | 9 | 11
Not completed — Death | 0 | 4
Not completed — Lack of Efficacy | 2 | 3
Not completed — Pregnancy | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 11 | 11
Not completed — Study Terminated by Sponsor | 76 | 120
Not completed — Other | 4 | 3
Not completed — Initiated prohibited medication | 0 | 2
Period: Open-label Extension Period: Week 52-113
Arm/Group | Placebo to Ustekinumab | Ustekinumab
Started | 88 | 137
Completed | 0 | 0
Not Completed | 88 | 137
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Study Terminated by Sponsor | 87 | 134

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo to Ustekinumab | Ustekinumab | Total
Number analyzed (Participants) | 208 | 308 | 516
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 1 | 4
  Between 18 and 65 years | 191 | 294 | 485
  >=65 years | 14 | 13 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (12.31) | 42.9 (11.38) | 43.5 (11.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 191 | 291 | 482
  Male | 17 | 17 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 45 | 79
  Not Hispanic or Latino | 172 | 263 | 435
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 7 | 9
  Asian | 46 | 57 | 103
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 18 | 24 | 42
  White | 136 | 208 | 344
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 5 | 10 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 15 | 13 | 28
  BULGARIA | 11 | 16 | 27
  CANADA | 0 | 2 | 2
  CHINA | 4 | 4 | 8
  COLOMBIA | 7 | 10 | 17
  GERMANY | 9 | 10 | 19
  HUNGARY | 3 | 11 | 14
  JAPAN | 21 | 25 | 46
  LITHUANIA | 10 | 11 | 21
  POLAND | 17 | 21 | 38
  PORTUGAL | 0 | 1 | 1
  RUSSIAN FEDERATION | 11 | 19 | 30
  SERBIA | 14 | 28 | 42
  SOUTH AFRICA | 4 | 8 | 12
  SOUTH KOREA | 0 | 5 | 5
  SPAIN | 4 | 6 | 10
  TAIWAN | 11 | 14 | 25
  THAILAND | 7 | 5 | 12
  UKRAINE | 8 | 22 | 30
  UNITED STATES | 52 | 77 | 129

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a Systemic Lupus Erythematosus Responder Index-4 (SRI-4) Composite Response at Week 52
Description: SRI-4 response:>=4-point reduction in SLEDAI-2K total score, no British Isles Lupus Assessment Group (BILAG) A (severe disease) and no more than 1 new BILAG B (moderate disease) domain score and no worsening (<10 % increase)from baseline in Physician's Global Assessment(PGA).SLEDAI measures disease activity in 9 organ systems,higher scores=more severe disease activity.Each organ system measured as either absent/present within last 30 days and weighted score across systems was utilized to calculate total SLEDAI score(range:0=no symptoms to 105=presence of all defined symptoms). Improvement is defined as reduction in SLEDAI score (BILAG) Index: assessing clinical signs, symptoms,or laboratory parameters related to SLE,divided into 9 domains. Each domain can range from A=new domain activity, B=worse domain activity, C=same domain activity, D=improving domain activity to E=absence of domain activity. PGA assesses disease activity on visual analogue scale from very well(0)-very poor(10).
Time Frame: Week 52
Population: The projected full analysis set (FAS) was defined as those participants (participants who received at least 1 dose [partial or complete,intravenous [IV] or subcutaneous [SC] of study agent) who should have had a given visit based upon their latest scheduled study visit. Participants were set to non-responders if they met treatment failure (TF) or had data missing.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Ustekinumab | Ustekinumab
Number analyzed (Participants) | 116 | 173
percentage of participants | 56.0 | 43.9
Statistical Analysis 1: Comparison: Placebo to Ustekinumab vs Ustekinumab; Test type: Superiority; p = 0.042, Regression, Logistic; Odds Ratio (OR) = 0.6, 95% CI 2-sided [0.4 to 1.0]

2. Secondary Outcome: Time to First Flare
Description: Time to flare is defined as the time (in days) post baseline when the first flare occurs. It was calculated with flare defined as either 1 or more BILAG A (severe disease activity) or 2 or more new BILAG B (moderate disease activity) domain scores relative to baseline. BILAG was defined as a measure of alterations or intensification to therapy consisting of 97 questions in 9 domains. Each domain can range from A=new domain activity, B=worse domain activity, C=same domain activity, D=improving domain activity to E=absence of domain activity. BILAG A flare was defined as at least 1 new BILAG A scores. BILAG B flare was defined as at least 2 new BILAG B scores.
Time Frame: Up to Week 52
Population: Analysis population is projected FAS. Participants were set to have flare if they met TF criteria (exceeded baseline dose of permitted SLE medications, initiated a new permitted SLE medication, initiated new protocol-prohibited medication or discontinued study agent for any reason prior to Week 52).
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo to Ustekinumab | Ustekinumab
Number analyzed (Participants) | 116 | 173
days
  Time to First BILAG Flare | 200.4 (121.27) | 204.7 (107.82)
  Time to First BILAG A Flare | 201.4 (122.83) | 203.1 (108.37)
  Time to First BILAG B Flare | 218.1 (125.00) | 208.7 (107.51)

3. Secondary Outcome: Percentage of Participants With an SRI-4 Composite Response at Week 24
Description: SRI-4 response:>=4-point reduction in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) total score, no BILAG A (severe disease) and no more than 1 new BILAG B (moderate disease) domain score and no worsening (<10 % increase)from baseline in PGA.SLEDAI measures disease activity in 9 organ systems, higher scores=more severe disease activity. Each organ system measured as either absent/present within last 30 days and weighted score across systems was utilized to calculate total SLEDAI score(range:0=no symptoms to 105=presence of all defined symptoms). Improvement is defined as reduction in SLEDAI score (BILAG) Index: assessing clinical signs, symptoms,or laboratory parameters related to SLE,divided into 9 domains. Each domain can range from A=new domain activity, B=worse domain activity, C=same domain activity, D=improving domain activity to E=absence of domain activity. PGA assesses disease activity on visual analogue scale from very well(0)-very poor(10).
Time Frame: Week 24
Population: Population analyzed included projected analysis set among participants who had or should have had a Week 24 visit based upon their last scheduled visit.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Ustekinumab | Ustekinumab
Number analyzed (Participants) | 116 | 173
percentage of participants | 56 | 45.7

4. Secondary Outcome: Percentage of Participants With 50 Percent (%) Improvement in Joints With Pain and Signs of Inflammation (Active Joints) at Week 52
Description: The percentage of participants who achieved at least 50% improvement from baseline in number of joints with pain and signs of inflammation at Week 52 for participants with at least 4 joints with pain and signs of inflammation at baseline were reported.
Time Frame: Week 52
Population: Analysis population is projected analysis set which included participants who had at least 4 joints with pain and signs of inflammation at baseline. Here, 'N' (number of participants analyzed) refers to participants evaluable included participants who had or should have had a Week 52 visit based upon their last scheduled visit and the date of trial termination.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Ustekinumab | Ustekinumab
Number analyzed (Participants) | 101 | 153
percentage of participants | 66.3 | 64.7

5. Secondary Outcome: Percentage of Participants Receiving Glucocorticoid at Baseline Who Achieved Change in Glucocorticoid Dose by Week 40 and Sustain That Change Through Week 52
Description: Reduction of glucocorticoid dose was defined as a reduction in average daily oral glucocorticoid dose by at least 50% (relative to the baseline dose) or reduction of average daily oral glucocorticoid dose by at least 25% (relative to the baseline dose) so that the average daily dose was reduced to less than or equal to (<=) 7.5 milligram (mg) (prednisone or equivalent). Sustained reduction of glucocorticoid dose was defined as achieving an average daily oral glucocorticoid dose reduction between Weeks 24 and 40, and sustaining that reduction through Week 52, in those participants who, at baseline, were receiving oral glucocorticoids.
Time Frame: Up to Week 52
Population: Analysis population is projected analysis set which included participants who received glucocorticoids at baseline. Here, 'N' (number of participants analyzed) refers to participants evaluable including participants who had or should have had a Week 52 visit based upon their last scheduled visit and the date of trial termination. Participants were set to non-responders if they met TF or had data missing.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Ustekinumab | Ustekinumab
Number analyzed (Participants) | 92 | 140
percentage of participants | 29.3 | 44.3

6. Secondary Outcome: Percentage of Participants With at Least a 50% Improvement in the Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) Activity Score at Week 52
Description: Percentage of participants achieving at least 50% improvement in CLASI activity score at Week 52 reported in participants with a CLASI activity score of 4 or greater at baseline. The CLASI is an instrument to assess the disease activity and damage caused to the skin for cutaneous lupus erythematosus participants with or without systemic involvement. The CLASI activity score ranges from 0-70 with lower score being improved. Activity is scored based on erythema, scale/hyperkeratosis, mucous membrane involvement, acute hair loss, and non-scarring alopecia.
Time Frame: Week 52
Population: Analysis population is projected FAS. Here, 'N' (number of participants analyzed) refers to participants who had or should have had a Week 52 visit based upon their last scheduled visit and the date of trial termination and with a CLASI activity score of 4 or greater at baseline. Participants were set to non-responders if they met TF or had data missing.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Ustekinumab | Ustekinumab
Number analyzed (Participants) | 93 | 135
percentage of participants | 55.9 | 40.7

7. Secondary Outcome: Percentage of Participants Receiving Glucocorticoid at Baseline Who Achieved Change in Glucocorticoid Dose by Week 40, Sustained That Change Through Week 52, and Achieved an SRI-4 Composite Response at Week 52
Description: Percentage of participants with reduction in glucocorticoid dose by Week 40, its sustenance through Week 52, and SRI 4 composite response at Week 52 were reported. Reduction of glucocorticoid dose was defined as reduction in average daily oral glucocorticoid dose by at least 50% (relative to baseline dose) or reduction of average daily oral glucocorticoid dose by at least 25% (relative to baseline dose) so that average daily dose is reduced to <=7.5 mg (prednisone or equivalent). Sustained reduction of glucocorticoid dose was defined as achieving an average daily oral glucocorticoid dose reduction between Weeks 24 and 40, and sustaining that reduction through Week 52, in those participants who,at baseline,were receiving oral glucocorticoids. SRI-4 was defined as composite of at least 4-point improvement in SLEDAI-2K score of 0=no symptoms to 105=presence of all defined symptoms with higher scores representing increased disease activity),no worsening in BILAG and no worsening in PGA.
Time Frame: Up to Week 52
Population: Analysis population is projected analysis set which included participants who received glucocorticoids at baseline. Here, 'N' (number of participants analyzed) refers to participants evaluable included participants who had or should have had a Week 52 visit based upon their last scheduled visit and the date of trial termination. Participants were set to non-responders if they met TF or had data missing.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Ustekinumab | Ustekinumab
Number analyzed (Participants) | 92 | 140
percentage of participants | 23.9 | 30.0

ADVERSE EVENTS:
Time Frame: Up to Week 130
Description: Safety analysis set included participants who were randomized, received at least 1 dose (partial or complete, intravenous or subcutaneous) of ustekinumab or placebo, and contributed any safety data after the start of study treatment. Participants received study drug up to Week 113, but were assessed for safety up to Week 130 (that is, after study termination). Participants were analyzed according to the actual treatment received.
Groups:
- Placebo (Prior to Entering (Long Term Extension [LTE]): Participants received matching placebo to ustekinumab intravenously (IV) 6 milligrams per kilogram (mg/kg) IV based on body weight at Week 0 followed by matching placebo to ustekinumab subcutaneously (SC) 90 mg at Week 8 and every 8 weeks (q8w) thereafter through Week 48 during double-blind period.
- Placebo to Ustekinumab (After Entering LTE): Participants who entered the open-label extension period at Week 52 crossed over to receive ustekinumab 90 mg SC q8w through Week 113.
- Ustekinumab (Through Week 113): Participants received ustekinumab 6 mg/kg IV based on body weight (ustekinumab 260 mg [weight less than or equal to (<=) 55 kg]; ustekinumab 390 mg [weight greater than {>} 55 kg and <= 85 kg] at Week 0 followed by ustekinumab 90 mg SC at Week 8 and q8w thereafter through Week 48 during double-blind period. At Week 52, participants who entered the extension period continued to receive ustekinumab 90 mg SC q8w through Week 113.
Arm/Group | Placebo (Prior to Entering (Long Term Extension [LTE]) | Placebo to Ustekinumab (After Entering LTE) | Ustekinumab (Through Week 113)
All-Cause Mortality (participants affected / at risk) | 1/208 | 0/88 | 5/307
Serious Adverse Events (participants affected / at risk) | 28/208 | 5/88 | 44/307
Other Adverse Events (participants affected / at risk) | 60/208 | 3/88 | 79/307
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Prior to Entering (Long Term Extension [LTE]) (N=208) | Placebo to Ustekinumab (After Entering LTE) (N=88) | Ustekinumab (Through Week 113) (N=307)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 2 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Cardiac Failure (Cardiac disorders) | 0 | 0 | 2
Pericardial Effusion (Cardiac disorders) | 0 | 0 | 1
Retinal Detachment (Eye disorders) | 1 | 0 | 0
Visual Impairment (Eye disorders) | 0 | 1 | 0
Abdominal Hernia (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Hepatorenal Syndrome (Hepatobiliary disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 4
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Endocarditis Staphylococcal (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 2
Herpes Zoster (Infections and infestations) | 1 | 0 | 0
Infected Bite (Infections and infestations) | 0 | 0 | 1
Nosocomial Infection (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 4
Pulmonary Tuberculosis (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 2 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 0
Viral Infection (Infections and infestations) | 1 | 0 | 0
Vulval Cellulitis (Infections and infestations) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Implantation Complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Patella Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post Procedural Fever (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Splenic Rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ulna Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Electrolyte Imbalance (Metabolism and nutrition disorders) | 1 | 0 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 4 | 0 | 2
Acoustic Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Diffuse Large B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Amnesia (Nervous system disorders) | 1 | 0 | 0
Embolic Stroke (Nervous system disorders) | 0 | 0 | 1
Facial Paralysis (Nervous system disorders) | 0 | 0 | 1
Haemorrhagic Stroke (Nervous system disorders) | 0 | 0 | 1
Neuropsychiatric Lupus (Nervous system disorders) | 0 | 0 | 2
Seizure (Nervous system disorders) | 0 | 0 | 1
Hyperemesis Gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0
Lupus Nephritis (Renal and urinary disorders) | 0 | 0 | 1
Nephritic Syndrome (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 2
Neurogenic Bladder (Renal and urinary disorders) | 1 | 0 | 0
Renal Colic (Renal and urinary disorders) | 0 | 0 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Ovarian Cyst (Reproductive system and breast disorders) | 0 | 0 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Lupus Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dermal Cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypersensitivity Vasculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Toxic Epidermal Necrolysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Aortic Aneurysm (Vascular disorders) | 0 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1
Hypovolaemic Shock (Vascular disorders) | 0 | 0 | 1
Lupus Vasculitis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Prior to Entering (Long Term Extension [LTE]) (N=208) | Placebo to Ustekinumab (After Entering LTE) (N=88) | Ustekinumab (Through Week 113) (N=307)
Nasopharyngitis (Infections and infestations) | 19 | 2 | 24
Upper Respiratory Tract Infection (Infections and infestations) | 17 | 0 | 25
Urinary Tract Infection (Infections and infestations) | 20 | 0 | 26
Headache (Nervous system disorders) | 14 | 1 | 19

LIMITATIONS AND CAVEATS:
Due to study termination, the open-label extension phase didn't reach the planned duration till Week 176. However, participants were assessed for safety up to Week 130 (that is, after study termination) and received study drug up to Week 113.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation.

DOCUMENTS (2):
  • Study Protocol (2019-01-23): https://cdn.clinicaltrials.gov/large-docs/22/NCT03517722/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-23): https://cdn.clinicaltrials.gov/large-docs/22/NCT03517722/SAP_001.pdf